CLINICAL TRIAL: NCT01582802
Title: Determinants of Neonatal Iron Homeostasis in Women Carrying Multiples
Brief Title: Determinants of Neonatal Anemia in Women Carrying Multiples
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: OSP 64155
Record Dates: First submitted 2012-04-12; First posted 2012-04-23 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal and cord blood, placental tissue and RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women carrying multiples: Healthy pregnant women carrying twins, triplets and quadruplets will be recruited.

SUMMARY:
Multiple births in the United States are rapidly increasing in large part due to assisted reproductive technologies. Recent data indicate that multiple births now comprise 3-4.5% of all births in the United States. Pregnant women are at risk for iron (Fe) deficiency anemia yet there are virtually no data on Fe status in women carrying multiples and current recommendations do not necessitate Fe screening among this high risk group. Maternal anemia is known to increase the risk of adverse birth outcomes including preterm birth and low birth weight. Moreover, the developing brain is increasingly recognized to be susceptible to Fe insufficiency in utero and growing data support that suboptimal Fe stores at birth are associated with long-term irreversible cognitive deficits in the offspring. To address these gaps in knowledge the investigators will monitor weight gain, hematological measures, Fe status indicators and serum hepcidin across pregnancy in approximately 120 women carrying twins and triplets. Determinants of maternal anemia will be identified. Neonatal hematological measures will be assessed in cord blood from each neonate at birth for assessment of hematological measures, Fe status and hepcidin. Determinants of neonatal anemia will be identified. Inflammatory markers will be measured in all blood samples and related to outcomes. Stable iron isotopes will be given to a subset of women to assess maternal Fe absorption and fetal Fe uptake.

DETAILED DESCRIPTION:
Pregnant women (n=100-125) carrying multiples (twins and triplets) will be identified when entering prenatal care. Women will be invited to participate in a longitudinal study of Fe homeostasis across pregnancy and at delivery in the maternal / neonatal dyad. In all maternal and cord blood samples obtained, whole blood will be analyzed for hemoglobin, hematocrit, reticulocyte count, erythrocyte count, mean corpuscular hemoglobin, mean corpuscular Hb concentration, mean corpuscular volume, and red cell distribution width using standard procedures. Circulating Fe status indicators (serum iron, ferritin, C-reactive protein, IL-6, erythropoietin, transferrin receptor and hepcidin) and serum folate and vitamin B12 will be measured. Distributions of each variable will be examined and associations among variables will be explored. Multiple linear regression models will be constructed to examine specific relations between a) determinants of Fe deficiency anemia in the mother; b) Fe status indicators in the mother vs. those in the neonate; c) Fe status indicators in the mother and neonate with placental Fe binding proteins; and d) neonatal Fe status between siblings.

ELIGIBILITY:
Inclusion Criteria:

* The investigators anticipate that the majority of these women will be recruited early in gestation because many of these pregnancies are a result of assisted reproductive technology.
* Eligible volunteers will be otherwise healthy and have no diagnosed, preexisting medical conditions known to impact iron homeostasis

Exclusion Criteria:

* Hemoglobinopathies,
* Preexisting diabetes,
* Malabsorption diseases

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women (n = 100-125) carrying multiples (twins, triplets and quadruplets)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-07; Primary Completion 2017-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Maternal iron status | Biochemical measures will be obtained whenever women have blood drawn across pregnancy (there are no fixed time points for sampling). These will be obtained over an approximate 36 week interval
  Maternal hematological measures will be evaluated
Neonatal iron status at birth | Umbilical cord blood will be collected at birth
  Cord blood hematological measures will be evaluated
Determinants of inter- and intra-uterine variance of neonatal iron status | Umbilical cord blood will be collected at birth
  ICC will be evaluated for iron status biomarkers

SECONDARY OUTCOMES:
Effect of maternal Fe status on placental iron transporter expression | Participants will be followed over the course of gestation from approximately week 12 of pregnancy until term
  protein and RNA expression of iron transporters will be evaluated
Maternal iron absorption and Fe57 enrichment in cord blood | Participants will be given 10 mg of stable iron between week 27-32 of gestation. Blood will be drawn 2 weeks post-dosing and maternal and umbilical cord blood will be obtained at delivery
  net quantity of isotope in newborns will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ru Y, Pressman EK, Cooper EM, Guillet R, Katzman PJ, Kent TR, Bacak SJ, O'Brien KO. Iron deficiency and anemia are prevalent in women with multiple gestations. Am J Clin Nutr. 2016 Oct;104(4):1052-1060. doi: 10.3945/ajcn.115.126284. Epub 2016 Aug 31. PMID 27581469
- [Background] Ru Y, Pressman EK, Guillet R, Katzman PJ, Bacak SJ, O'Brien KO. Predictors of anemia and iron status at birth in neonates born to women carrying multiple fetuses. Pediatr Res. 2018 Aug;84(2):199-204. doi: 10.1038/s41390-018-0044-6. Epub 2018 Jun 15. PMID 29907852
- [Background] Ru Y, Pressman EK, Guillet R, Katzman PJ, Vermeylen F, O'Brien KO. Umbilical Cord Hepcidin Concentrations Are Positively Associated with the Variance in Iron Status among Multiple Birth Neonates. J Nutr. 2018 Nov 1;148(11):1716-1722. doi: 10.1093/jn/nxy151. PMID 30247706
- [Derived] Barad A, Guillet R, Pressman EK, Katzman PJ, Ganz T, Nemeth E, O'Brien KO. Placental ferroportin protein abundance is associated with neonatal erythropoietic activity and iron status in newborns at high risk for iron deficiency and anemia. Am J Clin Nutr. 2024 Jan;119(1):76-86. doi: 10.1016/j.ajcnut.2023.10.022. Epub 2023 Oct 27. PMID 37890671
- [Derived] Delaney KM, Barad A, Castillo LF, Hasund CM, Guillet R, Pressman EK, Katzman PJ, Ganz T, Nemeth E, O'Brien KO. Placental Erythroferrone and Erythropoietin mRNA Expression is not Associated with Maternal or Neonatal Iron Status in Adolescents Carrying Singletons and Adult Women Carrying Multiples. J Nutr. 2023 Jul;153(7):1950-1958. doi: 10.1016/j.tjnut.2023.05.023. Epub 2023 May 28. PMID 37253412
- [Derived] Delaney KM, Guillet R, Pressman EK, Caulfield LE, Zavaleta N, Abrams SA, O'Brien KO. Iron absorption during pregnancy is underestimated when iron utilization by the placenta and fetus is ignored. Am J Clin Nutr. 2020 Sep 1;112(3):576-585. doi: 10.1093/ajcn/nqaa155. PMID 32614379
- [Derived] Delaney KM, Guillet R, Fleming RE, Ru Y, Pressman EK, Vermeylen F, Nemeth E, O'Brien KO. Umbilical Cord Serum Ferritin Concentration is Inversely Associated with Umbilical Cord Hemoglobin in Neonates Born to Adolescents Carrying Singletons and Women Carrying Multiples. J Nutr. 2019 Mar 1;149(3):406-415. doi: 10.1093/jn/nxy286. PMID 30770543